CLINICAL TRIAL: NCT04941339
Title: A Phase I, Open-label, Multi-center, First in Human, Dose Escalation and Expansion Study to Assess the Safety, Tolerability, Efficacy and Pharmacokinetics of MRG002 in Patients With HER2 Positive Advanced Solid Tumors
Brief Title: A Study of MRG002 in the Treatment of Patients With HER2-positive Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Miracogen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRG002-001
Record Dates: First submitted 2021-06-20; First posted 2021-06-28 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: Advanced Solid Tumor
Keywords: MRG002; Antibody Drug Conjugate (ADC); HER2; Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRG002 (Experimental): All patients in Phase Ia (dose escalation) and Phase Ib (dose expansion) will be administrated MRG002 on Day 1 of every 3 weeks (21-day cycle).
  Interventions: Drug: MRG002

INTERVENTIONS:
Drug: MRG002 — Administrated intravenously

SUMMARY:
The objective of this study is to assess the safety, efficacy, pharmacokinetics, and immunogenicity of MRG002 in patients with HER2-positive advanced solid tumors.

DETAILED DESCRIPTION:
This study consists of two parts. Phase Ia is a dose escalation study to determine the maximum tolerated dose (MTD) and recommended phase II dose (RP2D) of MRG002. Phase Ib is a dose expansion study to further assess the efficacy and safety of MRG002 at confirmed RP2D.

ELIGIBILITY:
Inclusion Criteria:

1. Understands and provides written informed consent and willing to follow the requirements specified in protocol;
2. Both genders;
3. Aged 18 to 75 (including 18 and 75);
4. Expected survival time ≥ 12 weeks;
5. Patients with histologically and/or cytologically confirmed HER2-positive solid tumors who have failed standard therapy or for whom no standard therapy exists or for whom standard therapy is not appropriate at current stage;
6. Patients must have at least one evaluable lesion (Phase Ia) or measurable lesion (Phase Ib) according to the Response Evaluation Criteria in Solid Tumors (RECIST 1.1);
7. The score of ECOG for performance status is 0 or 1;
8. Prior anti-tumor treatment-related AEs (NCI CTCAE v5.0 Criteria) have recovered to ≤ Grade 1 (except alopecia);
9. No severe cardiac dysfunction with left ventricular ejection fraction (LVEF) ≥ 50%;
10. Organ functions must meet the basic requirements;
11. Coagulation function must meet the basic requirements;
12. Cumulative anthracycline dose ≤ 360 mg/m2 doxorubicin or its equivalent, 720 mg/m2 epirubicin.

Exclusion Criteria:

1. Received radiotherapy, chemotherapy, biotherapy, immunotherapy, or other anti-tumor drugs within 3 weeks prior to the first dose of MRG002 treatment;
2. History of severe cardiac disease;
3. Clinically significant abnormalities in rhythm, conduction, and resting ECG morphology;
4. Patients with poorly controlled hypertension or clinically significant vascular disease;
5. History of moderate to severe dyspnea at rest due to advanced cancer or their complications, severe primary lung disease, or current need of continuous oxygen therapy, or any history of interstitial lung disease (ILD) or pneumonitis;
6. Nausea and vomiting of any kind difficult to control, or chronic gastrointestinal disease;
7. Patients with symptoms of central nervous system or brain metastasis or received treatment for central nervous system or brain metastasis within 3 months prior to the first dose of MRG002 treatment;
8. Major surgery not fully recovery within 4 months prior to the first dose of MRG002 treatment;
9. History of hypersensitivity to any component of MRG002 or history of hypersensitivity of ≥ Grade 3 to trastuzumab injection;
10. Evidence of active infection of hepatitis B or hepatitis C;
11. History of immunodeficiency, including human immunodeficiency virus (HIV) infection, or other immunodeficiency disease, or history of organ transplantation;
12. Any serious and/or uncontrolled disease or other condition that, considered by the investigator and sponsor, may compromise the patient's participation in this study;
13. Received systemic corticosteroids within 4 weeks prior to the first dose of MRG002 treatment;
14. Female patients with a positive serum pregnancy test or who are breast-feeding or who do not agree to take adequate contraceptive measures during the treatment and for 6 months after the last dose of study treatment.
15. Other conditions inappropriate for participation in this clinical trial, at the discretion of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2018-11-21 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | DLT will be evaluated during the first treatment cycle (Day 1-28)
  The highest dose confirmed wherein ≤ 1/6 of patients in a treatment cohort experiences a dose-limiting toxicity (DLT).
Recommended Phase II Dose (RP2D) | Baseline to study completion (up to 6 months)
  The dose level of MRG002 recommended for further clinical studies based on assessment of the safety, efficacy and PK data from this study.
Adverse Events (AEs) | Baseline to 49 days after the last dose of study treatment
  Any reaction, side effect, or untoward event that occurs during the course of the clinical trial whether or not the event is considered related to the study drug.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Baseline to study completion (up to 6 months)
  ORR is defined as the proportion of subjects with CR and PR assessed by IRC and investigator according to RECIST v1.1.
Duration of Response (DoR) | Baseline to study completion (up to 6 months)
  DoR is defined as the duration from the initial recording of objective disease response to the first onset of tumor progression, or death of any cause.
Progression Free Survival (PFS) | Baseline to study completion (up to 6 months)
  PFS is defined as the duration from the start of treatment to the onset of tumor progression or death of any cause.
Pharmacokinetics (PK) parameter of MRG002: Cmax | Baseline to 21 days after the last dose of study treatment
  Maximum observed plasma concentration.
Pharmacokinetics (PK) parameter of MRG002: Tmax | Baseline to 21 days after the last dose of study treatment
  Time to reach maximum plasma concentration.
Pharmacokinetics (PK) parameter of MRG002: t1/2 | Baseline to 21 days after the last dose of study treatment
  The time required for plasma concentration to decreased by on half.
Pharmacokinetics (PK) parameter of MRG002: AUClast | Baseline to 21 days after the last dose of study treatment
  Area under the curve up to the last validated measurable plasma concentration.
Immunogenicity | Baseline to 21 days after the last dose of study treatment
  The proportion of patients with positive ADA immunogenicity results.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, Doctor, Principal Investigator — Shanghai Oriental Hospital
Locations (1):
- Shanghai Oriental Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No